CLINICAL TRIAL: NCT01852396
Title: Ultrasound-Guided Brachial Plexus Regional Anesthesia by the Novel Retroclavicular Approach : A Feasibility Study
Brief Title: The Retroclavicular Approach for Regional Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Pablo Echave, Anesthesiologist, Université de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-020
Record Dates: First submitted 2013-04-22; First posted 2013-05-13 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Describe Novel Approach to Brachial Plexus Anesthesia
Keywords: Infraclavicular block; Brachial Plexus; Retroclavicular Approach; Complications of retroclavicular approach; Success of retroclavicular approach

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Regional anesthesia (Experimental): Recruit 50 patient having elbow, forearm, wrist or hand surgery and block brachial plexus using the novel retroclavicular approach
  Interventions: Procedure: Retroclavicular block

INTERVENTIONS:
Procedure: Retroclavicular block — Retroclavicular approach ultrasound guided regional anesthesia

SUMMARY:
The goal of this study is to demonstrate that the novel retroclavicular approach is a safe, fast and effective technique for ultrasound-guided brachial plexus anesthesia.

DETAILED DESCRIPTION:
Classic infraclavicular approach of the brachial plexus involves a needle puncture below the clavicle and advancing the needle with a 45-60 degree angle from cephalad to caudad. The aim is to advanced the block needle posterior to the axillary artery and to deposit the local anesthetic at that point, near the posterior cord. A "U" shaped spread around the artery should ensure distribution around all three cords. Ultrasound guidance is highly recommended and neurostimulation is optional.

The retroclavicular approach is a variant to this classical technique. Ultrasound probe is positioned initially below the clavicle in a manner similar to the classic approach but is then rotated in a clockwise fashion (right arm) or counter-clockwise fashion (left arm) for about 25-35 degrees. The puncture site is just behind the clavicle at the most lateral point available. If initial entry point is optimal, needle direction is then parallel to ultrasound probe. The final aim and position of block needle is identical to classical approach. Entry point ensures a parallel alignment of the needle and the ultrasound beam, thus enabling almost perfect visualization of both artery, cords and block needle. This is turn optimizes safety, rapidity of technique, efficiency and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Elective or Urgent Surgery of the hand, wrist or forearm
* 18 years and older
* Ability to consent
* American Society of Anesthesiologists class 1 to 3

Exclusion Criteria:

* Infection at the site of infection
* Abnormal anatomy at the site of infection
* Coagulopathy
* Severe Pulmonary Disease
* Preexisting neurological symptom(s) in the operated arm
* Pregnant patients
* Patients weighing less than 50 kg
* Allergy to amide type local anesthetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Success Rate of the Block | Assessed 30 minutes after block completion
  Success is defined as complete sensory loss in the distribution of the radial, median, ulnar, musculocutaneous, and medial cutaneous nerves of the forearm and hand.

SECONDARY OUTCOMES:
Surgical success rate | Defined at the beginning of surgery until the end of surgery
  Success rate is defined as avoidance of rescue analgesic technique. These techniques are defined as: adding local anesthetic locally by surgeon, rescue intravenous narcotics in excess of 1 microgram per kilogram of patient weight, need for general anesthesia, rescue distal neural blockage by anesthesiologist. Data presented will be the need or not of a rescue analgesic technique
Technique duration | Time required in seconds for the retroclavicular block technique completion, assessed during block performance
  Number of seconds needed to complete the block, from time of local skin anesthesia until regional block needle removal (local skin anesthesia plus injection of mepivacaine)
Needle visualization | Assessed after study completion, once all 50 patients will have been completed. Assessment will take place in the weeks following study completion
  Using the Likert standardized scale, two evaluators will individually quantify the ease of needle visualization using the video footage recorded by the ultrasound machine from all the retroclavicular blocks. Likert scale for visualization, is defined as: 1:very bad, 2: bad, 3: adequate, 4:good, 5: very good. No units are attached to this scale
Patient discomfort | Assessed immediately after the block
  Using a Visual Analog Scale (VAS), patients will quantify the discomfort they experienced during the block. This assessment will take place in the minutes following mepivacaine injection and block needle withdrawal. The VAS scale is rated from 1-10, 1 being almost no pain and 10 being the worst pain ever.
  Assessment will be done by an independent person, not taking part in the study. The VAS has no units attached to it.
Patient satisfaction | Assessed 48 hours after the block
  Using a VAS, patients will quantify their satisfaction with the retroclavicular technique throughout the study period.
Sensitive Block Progression | Assessed 10, 20, 30 minutes after the block
  Progress of the sensory block in the distribution of the radial, median, ulnar, musculocutaneous, and medial cutaneous nerves of the forearm and hand at 10, 20 and 30 minutes after block completion (mepivacaine injection). The scale used is: 0:no sensitive block, 1:analgesia, 2:anesthesia. No units are attached to this scale.
Motor Block Progression | Assessed 10, 20, 30 minutes after the block
  Progress of the motor block in the distribution of the radial, median, ulnar, musculocutaneous nerves of the forearm and hand at 10, 20, and 30 minutes after block completion (mepivacaine injection). The scale used is: 0: no motor block, 1: paresis, 2: paralysis. No units are attached to this scale
Complication Rate | Assessed 48 hours after the block
  With a phone call to the patient at 48 hours after injection of mepivacaine, complications will be searched for (pain at puncture site, paresthesia or paresis in the operated arm, signs of infection at puncture site such as redness or purulent discharge). Response is classified as YES or NO. No units attached to this scale. If patient reports paresthesia or paresis, further questioning over the phone will determine which nerve or cord is involved.
Duration of the Block's Effects | Assessed 48 hours after the block
  Duration of the block will be evaluated using 3 criteria: patient's subjective opinion of when the block receded (time of the day), time at which first oral analgesia is taken, and time of first onset of pain. Units involved is time (for example "3 pm".)
Use of narcotic for tourniquet pain | Assessed throughout the surgery
  If at any point during the surgery, patient complains of tourniquet pain, this will be noted as well as the analgesia given. Units is time of pain ("3 pm") and analgesia given ("micrograms of fentanyl").
Rate of Neurostimulation Usage | Assessed during the block
  At the discretion of the anesthesiologist performing the block, neurostimulation can be used to supplement ultrasound guidance. This will be recorded as a YES or NO (neurostimulation used or not). No units attached to this rate.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Echave, Doctor, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada